CLINICAL TRIAL: NCT00879866
Title: An Open-label, Phase Ib, Dose-escalation Trial on the Safety, Tolerability, Pharmacokinetics, Immunogenicity, Biological Effects and Antitumor Activity of EMD 521873 in Combination With Local Irradiation (20 Gy) of Primary Tumors or Metastases in Subjects With Non-small Cell Lung Cancer Stage IIIb With Malignant Pleural Effusion or Stage IV With Disease Control (Partial Response or Stable Disease) After Application of 4 Cycles of Platinum-based, First-line Chemotherapy
Brief Title: EMD 521873 Plus Radiotherapy in Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62235-002
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: NSCLC; immunocytokine; radiation; interleukin-2; immunotherapy; maintenance therapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — EMD 521873

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: EMD 521873

INTERVENTIONS:
Biological: EMD 521873 — After local irradiation (5 x 4 Gy) given over 5 consecutive days and 2 treatment free days cohorts of 3-6 subjects will receive EMD 521873 (as a 1h-infusion) on 3 consecutive days in 3-week cycles at dose levels of 0.15, 0.30, and 0.45 mg/kg, respectively.

SUMMARY:
Primary trial objective in this single arm trial is to assess the safety and tolerability of Selectikine (EMD 521873) given in combination with and local tumor irradiation and to determine whether the maximum tolerated dose (MTD) is reached with EMD 521873 doses of up to 0.45 mg/kg.

Secondary objectives are to evaluate PK, immunogenicity, overall response, changes in tumor marker levels and circulating tumor cell numbers, progression-free survival and overall survival. Also, to evaluate biological/immune responses to EMD 521873.

NSCLC patients have to be stable (PR or SD) after first-line chemotherapy in order to be enrolled. A total of 12 to 24 patients are planned. Patients will remain on the dose throughout the trial. It is intended to administer at least 4 cycles (21 d each), or until progression or 2nd line therapy becomes necessary.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC stage IIIb with malignant pleural effusion or stage IV
* Pulmonary primary tumor or at least one NSCLC metastasis in the lung measuring at least 1 cm in diameter and eligible for local radiation with 20 Gy
* Disease control (partial remission or stable disease) after 4 cycles of platinum-based first-line chemotherapy whereby the time between the last dose of first-line chemotherapy and start of trial treatment should not be longer than 8 weeks
* Male or female, aged ≥18 years of age
* Signed written informed consent
* Effective contraception for male and female subjects of childbearing age
* ECOG performance status 0 or 1
* Adequate hematological function defined by WBC ≥3 x 10^9/L, neutrophils ≥1.5 x 10^9/L, lymphocyte count ≥0.5 x 10^9/L, platelet count ≥100 x 10^9/L; hemoglobin ≥9 g/dL
* Estimated creatinine clearance ≥50 mL/min according to the Cockcroft - Gault formula or 24-h urine sampling
* Adequate hepatic function defined by a total bilirubin level ≤1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5 x ULN

Exclusion Criteria:

* Requirement for immunosuppressive treatment with the exception of inhalative corticosteroids or low-dose systemic corticosteroids (prednisone equivalent dose ≤10 mg/day)
* Systemic autoimmune disease (e.g. lupus erythematodes, rheumatoid arthritis)
* Organ transplant recipients
* Active infections (including HIV, hepatitis B and C, tuberculosis)
* Known or clinically suspected brain metastases
* Active cardiovascular/cerebrovascular disease (e.g. symptomatic coronary vascular disease, congestive heart failure ≥ NYHA II, LVEF <50%, ventricular arrhythmia requiring medication, myocardial infarction or stroke) within previous 6 months
* Pericardial effusion
* Major impairment in pulmonary function: forced expir¬atory volume in 1 second (FEV1) <50% and diffusion capacity for carbon monoxide (DLCO) <50% of normal limit
* Any other significant disease that in the Investigator's opinion would exclude the subject from the trial
* Known conditions associated with necroses of non-tumor bearing tissues (e.g. esophageal or gastroduodenal ulcers, ischemic bowel disease, chronic inflammations)
* Pregnancy or lactation
* Radiotherapy, chemotherapy, major surgery, biological therapy or any investigational drug within 30 days prior to the start of trial treatment
* Requirement for concurrent systemic anticancer treatment (chemotherapy, biological therapy)
* Pretreatment with anti-EGFR antibodies or tyrosine kinase inhibitors
* Participation in another interventional clinical trial within the past 30 days before start of trial treatment
* Known alcohol or drug abuse
* Any psychiatric condition that would prohibit the understanding or rendering of the informed consent
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of EMD 521873 given in combination with local irradiation of pulmonary primary tumor/metastases and to determine whether the maximum tolerated dose (MTD) is reached with EMD 521873 doses of up to 0.45 mg/kg. | Incidence of DLTs occurring during the first cycle (21 days) of administration of any dose of EMD 521873 following radiotherapy

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics (PK) of EMD 521873 in combination with local tumor irradiation | First 4 cycles of treatment
Evaluate the immunogenicity of EMD 521873 in combination with local tumor irradiation by measuring the induction of anti-EMD 521873 antibodies | First 4 cycles of treatment in each cycle, then every 4 cycles
Collect evidence of best overall response, changes in tumor marker levels and circulating tumor cell numbers after treatment with EMD 521873 in combination with local tumor irradiation | First 4 cycles of treatment
Collect evidence of best overall response after second-line therapy and duration of the response when it is shown | At one year of follow up
Evaluate progression-free survival and overall survival | At one year of follow up
Evaluate biological/immune responses following treatment with EMD 521873 by assessing changes in relevant parameters including leukocyte subset analysis | First 4 cycles of treatment
Evaluate biological/immune responses following treatment with EMD 521873 by assessing changes in relevant parameters including: molecular markers of immune activation (e.g. cytokines/chemokines, IL-2 receptor and neopterin) | First 4 cycles of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Quaratino, MD, PhD, Study Director — Merck KGaA, Darmstadt, Germany
Locations (3):
- Netherlands (3):
  - Department of Thoracic Oncology, Netherlands Cancer Instiute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Department of Pulmonology, Academic Hosptial Maastricht, Masstricht
  - Department of Medical Oncology (452), Radboud UMC Nijmegen, Nijmegen

REFERENCES:
- [Derived] Hendriks L, Dingemans AM, Lammens M, Anten MM, van den Heuvel MM, Postma LA. An Uncommon Presentation of Brain Metastases in a Lung Cancer Patient. J Thorac Oncol. 2015 Nov;10(11):1655-6. doi: 10.1097/JTO.0000000000000602. No abstract available. PMID 26536198
- [Derived] van den Heuvel MM, Verheij M, Boshuizen R, Belderbos J, Dingemans AM, De Ruysscher D, Laurent J, Tighe R, Haanen J, Quaratino S. NHS-IL2 combined with radiotherapy: preclinical rationale and phase Ib trial results in metastatic non-small cell lung cancer following first-line chemotherapy. J Transl Med. 2015 Jan 27;13:32. doi: 10.1186/s12967-015-0397-0. PMID 25622640